CLINICAL TRIAL: NCT05918133
Title: A Phase Ib/II Study of PM8002 Injection Plus Nab-paclitaxel as First Line Therapy for Unresectable, Locally Advanced or Metastatic Triple-negative Breast Cancer
Brief Title: A Study of PM8002 Plus Nab-paclitaxel as First Line Therapy for TNBC
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Biotheus Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PM8002-B004C-TNBC-R
Record Dates: First submitted 2023-06-15; First posted 2023-06-26 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2024-11

CONDITIONS: TNBC
Keywords: First line
MeSH Terms: interventions — 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PM8002+nab-paclitaxel (Other): PM8002 at 20 mg/kg (Q2W) and nab-paclitaxel at 100 mg/m2 on the 1st, 8th, and 15th days of each cycle until unacceptable toxicity or disease progression were observed. Each cycle contains 28 days.
  Interventions: Drug: PM8002; Drug: nab-paclitaxel

INTERVENTIONS:
Drug: PM8002 — IV infusion
Drug: nab-paclitaxel — IV infusion

SUMMARY:
Here, the investigators present the results from a Phase Ib/II study of PM8002 in combination with nab-paclitaxel in subjects with locally advanced or metastatic triple negative breast cancer without previous systematic treatment.

DETAILED DESCRIPTION:
PD-L1 and VEGF play important roles in immune escape and tumor angiogenesis and enhance cancer growth and metastasis. PM8002 is a bispecific antibody targeting PD-L1 and VEGF-A. Here, the investigators present the results from a Phase Ib/II study of PM8002 in combination with nab-paclitaxel in subjects with locally advanced or metastatic triple negative breast cancer without previous systematic treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily participate in clinical research; fully understand the study and voluntarily sign the informed consent; willing to follow and have the ability to complete all trial procedures;
2. Male or female, aged 18 to 75 years (including boundary value);
3. Unresectable locally advanced or metastatic breast cancer confirmed by histology or cytology, ER, PR, HER-2 are all negative. Negative ER and PR were defined as: IHCER < 1%, IHCPR < 1%. HER-2 negative is defined as: IHCHER-2 (-) or (1+), HER-2 (2+) must be tested by FISH and the result is negative.
4. Patients who have not received systemic treatment for advanced TNBC in the past are allowed to use taxane anti-tumor therapy in the previous neoadjuvant and/or adjuvant treatment stage, but must meet the end time of taxane neoadjuvant and/or adjuvant treatment Recurrence/metastasis interval ≥ 12 months;
5. Sufficient organ function;
6. The Eastern Cooperative Oncology Group (ECOG) score of physical status is 0-1;
7. Expected survival period ≥ 12 weeks;
8. According to the RECIST1.1 standard, the subject has at least one measurable tumor lesion.

Exclusion Criteria:

1. History of severe allergic diseases, allergic history of serious drugs (including unlisted test drugs) or known allergic to any component of this test drug;
2. Previously received any antibody or inhibitor therapy targeting PD-1/PD-L1 or VEGF;
3. There is meningeal metastasis, uncontrollable or symptomatic central nervous system (CNS) metastasis;
4. Those who have active infection and currently need intravenous anti-infection treatment;
5. At present, there are uncontrollable pleural effusion, pericardium effusion and abdominal effusion;
6. Before the start of the study and treatment, fever of unknown cause > 38.5°C (according to the researcher's judgment, fever caused by tumor can be included in the group);
7. Known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation;
8. Known history of alcohol abuse, psychotropic substance abuse or drug abuse;
9. Have a clear history of neurological or mental disorders, such as epilepsy, dementia and schizophrenia;
10. Human immunodeficiency virus (HIV) infection or known acquired immunodeficiency syndrome (AIDS);
11. Syphilis nonspecific antibody test is positive (such as TRUST and PRP) or syphilis specific antibody test is positive (such as TPPA) [it is acceptable that "Syphilis specific antibody test" is positive but "Syphilis nonspecific antibody test" is negative for more than one year];
12. Active tuberculosis, or a history of tuberculosis infection in the past but failed to control after treatment;
13. Active hepatitis B (HBsAg positive and HBV-DNA ≥1 1000 IU/ml) can be controlled by antiviral drugs (HBV-DNA < 1000 IU/ml). Active hepatitis C (HCV-RNA > detection limit of research center);
14. According to the researcher's judgment, the subject's basic illness may increase the risk of receiving the study drug, or confuse the explanation of the toxic reaction and AE;
15. It is expected that any other form of anti-tumor drug treatment will be required during the study;
16. Women who are pregnant or breastfeeding.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2026-10-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | Up to approximately 2 years
  Objective response rate (ORR) is the proportion of subjects with complete response (CR) or partial response (PR), based on RECIST v1.1
Treatment related adverse events (TRAEs) | Up to 30 days after last treatment]
  The incidence and severity of TRAEs graded according to NCI-CTCAE v5.0

SECONDARY OUTCOMES:
Disease control rate (DCR) | Up to approximately 2 years
  DCR is defined as the proportion of subjects with CR, PR, or stable disease(SD) based on RECIST v1.1.
Duration of response (DoR) | Up to approximately 2 years
  DoR is defined as the duration from the first documentation of objective response to the first documented disease progression (based on RECIST v1.1) or death due to any cause, whichever occurs first.
Progression free survival (PFS) | : Up to approximately 2 years
  PFS is defined as the time from the start of treatment until the first documentation of disease progression or death due to any cause, whichever occurs first (based on RECIST v1.1).
Overall survival (OS) | Up to approximately 2 years
  OS is the time from the date of first dosing date to death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Wu Jiong, Principal Investigator — Fudan University
Locations (8):
- China (8):
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Affiliated Cancer Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Nanchang Third Hospital, Nanchang, Jiangxi
  - The first ward of breast Surgery, Shandong Cancer Hospital, Jinan, Shandong
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Yibin Second People's Hospital, Yibin, Sichuan
  - Tian Jin Medicial University Cancer Institute&Hospital, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: Yes
The data will be published or presented for publications (poster, abstract,articles or papers) or any presentations.
Time Frame: After the trial completed.
Access Criteria: NCI is committed to sharing data in accordance with NIH policy.